CLINICAL TRIAL: NCT07030257
Title: A Multi-Center, Open Label, Phase 1/2 Study of CP-383, in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Study of CP-383 in Patients With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tasca Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAS-CP383-01
Record Dates: First submitted 2025-05-20; First posted 2025-06-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor Malignancies; Colorectal Carcinoma; Small Cell Lung Cancer ( SCLC ); Head and Neck (HNSCC); Bladder Cancer; Non-Small Cell Lung Cancer; Pancreatic Cancer, Advanced or Metastatic
Keywords: Phase 1; Dose Escalation; Dose Expansion; Loss of Function; FAT1; P300
MeSH Terms: conditions — Colorectal Neoplasms; Small Cell Lung Carcinoma; Squamous Cell Carcinoma of Head and Neck; Urinary Bladder Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Dose Level 1 (Experimental): CP-383, single daily oral capsule, 0.8 mg
  Interventions: Drug: CP-383
- Dose Level 2 (Experimental): CP-383, single daily oral capsule, 1.6 mg
  Interventions: Drug: CP-383
- Dose Level 3 (Experimental): CP-383, single daily oral capsule, 3.0 mg
  Interventions: Drug: CP-383
- Dose Level 4 (Experimental): CP-383, single daily oral capsule, 5.0 mg
  Interventions: Drug: CP-383
- Dose Level 5 (Experimental): CP-383, single daily oral capsule, 8.0 mg
  Interventions: Drug: CP-383
- Dose Level 6 (Experimental): CP-383, single daily oral capsule, 12 mg
  Interventions: Drug: CP-383
- Expansion Arm 1 (Experimental): Expansion in selected tumor type at recommended Phase 2 Dose of CP-383
  Interventions: Drug: CP-383
- Expansion Arm 2 (Experimental): Expansion in selected tumor type at recommended Phase 2 Dose of CP-383
  Interventions: Drug: CP-383
- Expansion Arm 3 (Experimental): Expansion in selected tumor type at recommended Phase 2 Dose of CP-383
  Interventions: Drug: CP-383
- Expansion Arm 4 (Experimental): Expansion in selected tumor type at recommended Phase 2 Dose of CP-383
  Interventions: Drug: CP-383

INTERVENTIONS:
Drug: CP-383 — Novel anti-cancer agent inhibiting pyrimidine synthesis in cancer cells

SUMMARY:
The goal of this clinical trial is to learn if an investigational drug CP-383 works to treat advanced cancer. It will also learn about the safety of CP-383. The main questions if aims to answer are:

* Does CP-383 slow or stop the growth of cancer in patients with advanced cancer
* What medical problems do participants have when taking CP-383 Researchers will test CP-383 in all kinds of cancers at various dose levels to determine what the best dose is to study further. Researchers will also see if certain cancers that have gene mutations respond better to CP-383

Participants will:

* Take CP-383 every day by mouth until the researcher learns whether CP-383 is helping slow or reduce the cancer growth
* Visit the clinic weekly for the first 6 weeks for checkups and tests
* Visit the clinic every 3 weeks thereafter for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Measurable or non measurable cancer that the research can assess for changes
* Not eligible or able to take existing standard therapies for cancer
* Availability of a part of a tumor for laboratory testing or willing to have a safe biopsy taken from a tumor
* Diagnosed with locally advanced, recurrent or metastatic incurable disease
* Part 1: any solid tumor (with the exception of brain cancer) that has progressed, standard therapy is no longer or has not helped the cancer, or is too toxic and for whom a clinical trial is an option for continued treatment
* Part 1: specific advanced, metastatic tumor types will also be enrolled: colorectal cancer, small cell lung cancer, head and neck cancer, non-small cell lung cancer, pancreatic cancer, bladder cancer - some of these will have a specific gene mutation in the cancer
* Part 1: selected solid tumor cancer types (with the exception of brain cancers) that have a specific gene mutation in the cancer
* Part 2: specific advanced, metastatic tumor types will also be enrolled: colorectal cancer, small cell lung cancer, head and neck cancer - some of these will have a specific gene mutation in the cancer

  _ Part 2: selected solid tumor cancer types (with the exception of brain cancers) that have a specific gene mutation in the cancer
* Adequate blood and urine lab tests
* Women and men of childbearing potential with adequate contraception
* Provides written informed consent
* Willing to comply with the requirements of the protocol

Exclusion Criteria:

* Inability to swallow pills
* Known history of HIV, HCV, HBV unless cured, controlled with undetectable viral load
* Active tumor in the brain
* Clinically significant liver disease
* Significant gastrointestinal diseases
* History of other cancer within past 5 years with certain exceptions for cancers that are likely cured
* Significant cardiac disease
* Other diseases that are not well controlled that could make taking the drug unsafe
* pregnant or lactating females
* Exposure to certain anti-cancer or other drugs within a certain period before the start of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2028-08-15 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Part 1: Determine the maximum tolerated dose (MTD) | 21 days
  Determine the MTD of CP-383 in subjects with advanced solid tumors
Part 2: Evaluate the efficacy of CP-383 at the recommended phase 2 dose in selected tumor types | From enrollment through study completion, an average of 1 year
  Objective response rate assessed by the investigator according to RECIST

SECONDARY OUTCOMES:
Part 1: Determine the pharmacokinetics parameters of CP-383 | From enrollment through study completion, an average of 1 year
  Assess standard PK parameters including Cmax
Part 1: Determine the pharmacokinetics parameters of CP-383 | From enrollment through study completion, an average of 1 year
  Assess standard PK parameters including tmax
Part 1: Determine the pharmacokinetics parameters of CP-383 | From enrollment through study completion, an average of 1 year
  Assess standard PK parameters including AUC
Part 1: Assess safety and tolerability of CP-383 in participants with advanced solid tumors | From enrollment through study completion, an average of 1 year
  Incidence and severity of Adverse events and changes in test results
Part 2: Evaluate safety and tolerability of CP-383 at the recommended Phase 2 dose in selected tumor types | From enrollment through study completion, an average of 1 year
  Incidence of AEs and changes in test results
Part 2: Evaluate the efficacy of CP-383 at the recommended phase 2 dose in selected tumor types | From enrollment through study completion, an average of 1 year
  Evaluate duration of response
Part 2: Evaluate the efficacy of CP-383 at the recommended phase 2 dose in selected tumor types | From enrollment through study completion, an average of 1 year
  Evaluate disease control as determined by Objective response of CR, PR or SD for at least 6 months
Part 2: Evaluate the efficacy of CP-383 at the recommended phase 2 dose in selected tumor types | From enrollment through study completion, an average of 1 year
  Evaluate progression free survival
Part 2: Evaluate the efficacy of CP-383 at the recommended phase 2 dose in selected tumor types | From enrollment through study completion, an average of 1 year
  Evaluate overall survival

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Florida Cancer Specialists-Lake Nona, Orlando, Florida
  - START Midwest, Grand Rapids, Michigan
  - Washington University, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Taylor Cancer Research Center, Maumee, Ohio
  - NEXT Oncology - Dallas, Dallas, Texas
  - START San Antonio, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Undecided